CLINICAL TRIAL: NCT06954831
Title: Phase 2 Trial of Ultra-Hypofractionated Whole Breast Irradiation With Concomitant Lumpectomy Cavity Boost
Brief Title: Ultra-hypofractionated Whole Breast Irradiation With Lumpectomy Cavity Boost for the Treatment of Stage I-III Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23860; NCI-2025-02185 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23860 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-05-02 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (UF-WBI with CB) (Experimental): Patients undergo UF-WBI with CB QD on consecutive business days for up to 5 fractions in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CBCT prior to each radiation treatment.
  Interventions: Procedure: Cone-Beam Computed Tomography; Radiation: Hypofractionated External Beam Radiation Therapy; Other: Questionnaire Administration; Radiation: Radiation Boost; Radiation: Whole Breast Irradiation

INTERVENTIONS:
Procedure: Cone-Beam Computed Tomography — Undergo CBCT
  Other Names: Cone Beam Computed Tomography; Cone Beam CT
Radiation: Hypofractionated External Beam Radiation Therapy — Undergo UF-WBI with CB
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Boost — Undergo UF-WBI with CB
  Other Names: BOOST; Boost Radiation; Boost Radiation Therapy; Boost Radiotherapy; Radiation Therapy Boost; Radiotherapy Boost
Radiation: Whole Breast Irradiation — Undergo UF-WBI with CB

SUMMARY:
This clinical trial tests how well ultra-hypofractionated (UF) whole breast irradiation (WBI) with lumpectomy cavity boost (CB) works in treating patients with stage I-III breast cancer. Breast conservation therapy (BCT) is the recommended treatment for patients with early stage breast cancer. BCT involves a lumpectomy followed by breast radiation. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Traditionally, WBI has been given once daily over 5-6 weeks and then those at high-risk for recurrence receive additional radiation (boost) to the lumpectomy cavity daily over 4-8 days. This has now been replaced by moderate hypofractionated radiation. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Although moderate hypofractionated radiation therapy reduces the length of treatment from 6-7 weeks to 3-4 weeks, the length of treatment still remains a barrier for many patients. UF-WBI with CB delivers radiation to the whole breast and the surgical cavity at the same time over 5 daily treatments. Giving UF-WBI with CB may prevent recurrence and prolong survival as well as improve the quality of life in patients with stage I-III breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the impact of UF-WBI + CB as assessed by patient-reported Global Cosmesis Score (GCS) at 1 year.

SECONDARY OBJECTIVES:

I. To characterize the patient-reported cosmetic appearance of the breast over time, as assessed by GCS.

II. To determine short- and long-term physician-reported cosmetic appearance of the breast, as assessed by GCS.

III. To evaluate the acute and late patient-reported radiation-associated toxicities.

IV. To evaluate the acute and late physician-reported radiation-associated toxicities.

V. To estimate:

Va. 5-year in-breast recurrence; Vb. 5-year distant recurrence; Vc. 5-year disease-free survival (DFS); Vd. 5-year overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To evaluate patient-reported quality-of-life (QoL). II. To evaluate volumetric and dosimetric factors associated with acceptable breast cosmesis.

III. To evaluate volumetric and dosimetric factors associated with acute and late radiation-associated toxicities.

OUTLINE:

Patients undergo UF-WBI with CB once daily (QD) on consecutive business days for up to 5 fractions in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo cone-beam computed tomography (CBCT) prior to each radiation treatment.

After completion of study treatment, patients are followed up at 1 month, 6 months, then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: ≥ 40 years
* Female
* Ability to read and understand English for questionnaires
* Histologically confirmed breast cancer
* Malignancy must be epithelial. Non-epithelial breast malignancies such as lymphoma or sarcoma are not allowed
* Patients must have undergone breast conserving surgery. Re-excision for negative margins is allowed
* Patients must have undergone surgical staging of the axilla (sentinel lymph node biopsy or axillary lymph node dissection)
* Must have at least one-high risk feature that would necessitate a lumpectomy cavity boost by the treating radiation oncologist
* Patient must have physician-reported "Excellent" or "Good" cosmesis post-lumpectomy and prior to radiation therapy based on the 4-point Global Cosmetic Score
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior radiation to the region of the involved breast that in the opinion of the investigator would preclude breast irradiation
* Pathologically or clinically involved regional lymph nodes necessitating comprehensive regional nodal irradiation that includes the supraclavicular fossa
* Clinically significant uncontrolled illness
* Stage IV breast cancer
* Diagnosis of Paget's disease of the nipple
* Other prior or active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Pregnant or breastfeeding
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | At 1 year
  Responding patients are defined as patients with a rating of either "excellent" or "good" on the 4-point Global Cosmesis Score (GCS). Will be estimated along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Patient-reported cosmetic outcome using GCS - Baseline | At baseline
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided.
Patient-reported cosmetic outcome using GCS - 6 months | At 6 months
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided.
Patient-reported cosmetic outcome using GCS - 1 year | At 1 year
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided.
Patient-reported cosmetic outcome using GCS - 2 years | At 2 years
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided.
Patient-reported cosmetic outcome using GCS - 3 years | At 3 years
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided.
Physician-reported cosmetic outcome using GCS | At baseline, at 6 months and at years 1, 2, and 3
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided.
Patient-reported radiation-associated toxicities | At 1 month, 6 months, and 1 year
  Will be assessed and graded using Patient-Reported Outcome Common Terminology Criteria for Adverse Events. Observed toxicities will be summarized by type, severity, and attribution. For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided.
Physician-reported radiation-associated toxicities | At 1 month, 6 months, and years 1, 2, and 3
  Will be assessed and graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Observed toxicities will be summarized by type, severity, and attribution. For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided.
Incidence of in-breast disease recurrence | Up to 5 years
  Will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided.
Incidence of metastatic disease | Up to 5 years
  Will be evaluated using RECIST criteria. For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided.
Disease free survival | From start of treatment to in-breast recurrence, metastatic disease, or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method with Greenwood variance estimator and 95% confidence interval will be constructed based on log-log transformation.
Overall survival | From start of treatment to death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method with Greenwood variance estimator and 95% confidence interval will be constructed based on log-log transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M Yoon, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (7):
- United States (7):
  - City of Hope at Arcadia, Arcadia, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope at South Bay, Torrance, California
  - City of Hope Upland, Upland, California